CLINICAL TRIAL: NCT02525120
Title: Post Market Non-Inferiority Study Comparing Triojection® to Discectomy for Lumbar Disc Herniation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minimus Spine, Inc (Other)
Collaborators: genae international,ag (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1CP-1
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Lumbar Disc Herniation
Keywords: Disc herniation; Herniated disc; Triojection; Ozone; Lumbar spine; Leg pain
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triojection System for ozone injection (Experimental): Triojection is a system including a single-use sterile syringe cartridge and an accessory console. The console is interfaced to a supply of medical oxygen and uses this supply to fill the syringe with oxygen. Ozone is produced by applying a high voltage to electrodes physically located within the syringe. When a concentration of 35µg/ml is reached, the cartridge is removed from the console. The sterile syringe, containing the gas, is extracted from the protective housing and the gas is administered directly to the center of the herniated disc through a spinal needle.
  Interventions: Device: Triojection
- Surgical discectomy (Active Comparator): The surgical group will be receive a standard surgical discectomy to remove the herniated disc material.
  Interventions: Procedure: Surgical discectomy

INTERVENTIONS:
Device: Triojection — Triojection is system intended to deliver a specific amount of ozone to a herniated disc.
  Arms: Triojection System for ozone injection
Procedure: Surgical discectomy — Patients will receive surgery to remove the herniated disc material.
  Arms: Surgical discectomy

SUMMARY:
The primary objective of this study is to compare the early clinical outcomes following non-surgical treatment with Triojection® to surgical discectomy. Early is defined as less than or equal to 6 months.

DETAILED DESCRIPTION:
The objective of this study is to compare clinical, economic and safety outcomes between Triojection and surgical discectomy. The study will include two follow-up phases: 1) an initial follow-up period during the first 6 months after treatment and (2) a long-term follow-up lasting an additional 18 months (2 years total).

The hypothesis is that over the first six months after treatment, Triojection® will be non-inferior to discectomy with respect to the improvement in leg pain. This will be demonstrated using a non-inferiority margin of 19.4 points on the difference between baseline leg pain score and the average leg pain score recorded at 1 week, 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria

1. Patient is willing to provide informed consent.
2. Clinical and radiographic evidence of one, and only one, symptomatic protruding or extruded disc between L1 and S1.
3. The herniated disc should have a disc height of at least 50% that of the normal adjacent disc levels, as determined by the investigator.
4. The signal intensity of the herniated disc material should be equal or greater than the nucleus pulposus of the herniated disc.
5. The patient must have pain in a dermatomal distribution consistent with their radiographic findings
6. Leg pain greater than or equal to 5 on the NRS scale
7. Symptoms for at least 6 weeks
8. Willingness to complete all follow-up evaluations
9. Patient aged 18-65 years
10. BMI<40

Exclusion Criteria:

1. Patients with a disc herniation extending past the facet joint
2. Presence of a non-contiguous disc fragment
3. Impairment of bladder/bowel function or motor impairment in the affected leg
4. An epidural steroid injection in the past 2 weeks
5. Previous discectomy, arthroplasty or fusion at any lumbar level
6. In patients with L5-S1 disc herniation, a congenital condition where the L5 vertebral body is either fused to the sacrum or the L5-S1 disc is not fully formed as a normal adult disc.
7. Symptomatic lumbar stenosis or listhesis
8. Symptomatic sacroiliac joint
9. Symptomatic foraminal stenosis due to severe degenerative disc disease
10. History of spinal tumor, fracture or infection
11. Females of childbearing age that are known to be pregnant or wishing to become pregnant during the study
12. Fibromyalgia
13. Active infection
14. Metastatic cancer within the past 5 years
15. Pending litigation against a health care provider
16. More than 3 months of continuous sick leave prior to enrollment.
17. Known drug or alcohol abuse
18. Diagnosed psychiatric disease or psychological distress caused by recent trauma like divorce, death of a member family or loss of a job
19. Patient known to be affected by favism (G6PD deficiency)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Leg pain NRS | Baseline, 1 week, 1, 3 and 6 months.
  The primary outcome measure will be the amount of improvement in leg pain after treatment. This will be determined by taking the difference between the baseline score and the average of the post-treatment scores at 1 week, 1, 3 and 6 months.

SECONDARY OUTCOMES:
Leg pain NRS | Baseline and 1 week, 1, 3, 6, 12, 18 and 24 months after treatment.
  Leg pain Numerical Rating Scale (NRS) at each visit.
Back pain NRS | Baseline and 1 week, 1, 3, 6, 12, 18 and 24 months after treatment.
  Back pain Numerical Rating Scale (NRS) at each visit
Functional Score measured by RMDI. | Baseline and 1 week, 1, 3, 6, 12, 18 and 24 months after treatment.
  Roland Morris Disability Index. A 24 question survey asking the subject if they have difficulty with various activities of daily living.
Quality of Life measured by EQ-5D | Baseline and 1 week, 1, 3, 6, 12, 18 and 24 months after treatment.
  EQ-5D is a validated survey asking the subject 5 multiple choice questions and to indicate their general health status on a scale of 0-100.
Patient Satisfaction via a survey | Baseline and 1 week, 1, 3, 6, 12, 18 and 24 months after treatment.
  Brief questionnaire asking patients to rate their level of satisfaction.
Cost Diary | Baseline and 1 week, 1, 3, 6, 12, 18 and 24 months after treatment.
  Survey asking patients to detail their medical expenses, work status, time off work etc.
Review of MRI images | Baseline and 6 and 24 months after treatment.
  Blinded, independent MRI review to determine reduction in disc herniation following treatment and evaluate index and adjacent levels for evidence of degeneration.

OTHER OUTCOMES:
Adverse Events | Through 24 months
  All adverse events are to be reported, per ISO 14155.

CONTACTS AND LOCATIONS:
Overall Officials: Josip Buric, MD, Study Director — Centro Chirurgico San Paolo, Pistoia, Italy
Locations (3):
- University General Hospital Attikon, Athens, Haidari, Greece
- Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Lombardy, Italy
- Ospedale Regionale di Lugano- Civico e Italiano, Lugano, Switzerland